CLINICAL TRIAL: NCT02156999
Title: Changes of Bone Turnover Markers and Bone Mineral Density After Treatment in Osteoporotic Patients
Brief Title: Changes of Bone Turnover Markers and Bone Mineral Density After Osteoporosis Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Assistant professor, Shinshu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2014
Record Dates: First submitted 2014-06-01; First posted 2014-06-05 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Osteoporosis (Experimental)
  Interventions: Device: Ibandronic acid, vitamin D

INTERVENTIONS:
Device: Ibandronic acid, vitamin D

SUMMARY:
To examine the changes of bone mineral density and bone turnover markers after Bonviva treatment in osteoporotic patients

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis

Exclusion Criteria:

* Kidney, parathyroid, congenital bone metabolic disease

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes of bone mineral density | every 4-6 months
  To examine the changes of bone mineral density for the purpose of the effectiveness of the drug

SECONDARY OUTCOMES:
Improvement of bone turnover markers | Every 3-6 months
  To examine the changes of bone turnover markers for the purpose of the effectiveness of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan